CLINICAL TRIAL: NCT04170439
Title: The Added Value of n Acetyle Cysteine and Chromium to Clomiphene Citrate in PCO
Brief Title: Added Value of N Acetyle Cysteine to Clomiphene Citrate in PCO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aljazeera Hospital (Other)
Collaborators: Cairo University (Other)
Responsible Party: Principal Investigator, Mahmoud Alalfy, Lecturer in national research crntre and Algezzera hospital ,egypt, Aljazeera Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: chromium in infertility
Record Dates: First submitted 2019-11-16; First posted 2019-11-20 (Actual); Last update posted 2021-04-28 (Actual); Status verified 2021-04

CONDITIONS: PCO
MeSH Terms: interventions — Clomiphene; Metformin; Chromium

STUDY DESIGN:
Intervention Model Description: Women who will receive clomiphe citrate plus N acetyle cysteine rally in arm number 1 And women who will receive clomiphene citrate and chromoum in arm number 22
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- clomiphene plus metformin plus N acetyle cysteine (Other): Women who will receive clomiphene citrate plus metformin plus n acetyle cysteine
  Interventions: Drug: Clomiphene plus metformin plus N acetyle cysteine in arm number 1
- clomiphene plus metformin plus chromium (Other): Women who will receive clomiphene plus metformin plus chromium
  Interventions: Drug: Clomiphene citrate plus metformin with chromium
- clomiphen citrate plus metformin (Other): Women who will receive clomiphene plus metformin
  Interventions: Drug: clomiphene citrate plus metformin

INTERVENTIONS:
Drug: Clomiphene plus metformin plus N acetyle cysteine in arm number 1 — oral adminstration of clomiphene citrate plus metformin plus N acetyl cysteine or chromium
  Arms: clomiphene plus metformin plus N acetyle cysteine
Drug: Clomiphene citrate plus metformin with chromium — oral adminstration of clomiphene citrate plus metformin and chromium
  Arms: clomiphene plus metformin plus chromium
Drug: clomiphene citrate plus metformin — oral adminstration of clomiphene citrate plus metformin
  Arms: clomiphen citrate plus metformin

SUMMARY:
PCO is one of the factors associated with delayed conception

DETAILED DESCRIPTION:
In an attempt to induce ovulation Clomiphene citrate can be given in conjunction with N acetyle cysteine

ELIGIBILITY:
Inclusion Criteria:

* women with PCO

Exclusion Criteria:

* women who donot have PCO

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Women with PCO
Enrollment: 108 (Actual)
Dates: Start 2019-11-20 (Actual); Primary Completion 2020-05-02 (Actual); Study Completion 2020-05-15 (Actual)

PRIMARY OUTCOMES:
The number of women who will have mature follicles wih their size and number of mqture follicles The number of women who will have mature follicles | within 2 weeks
  Assessment of women in both groups for size and number of follicles

CONTACTS AND LOCATIONS:
Overall Officials: Mahmoud Alalfy, PhD, Study Director — Algezeera
Locations (2):
- Egypt (2):
  - Algazeerah and Kasralainy hospital, Giza
  - Algazeerah, Giza